CLINICAL TRIAL: NCT04145908
Title: Non Absorbable Mesh Reinforcement of Midline Incision Closure in High Risk Patients, Onlay Versus Preperitoneal Position, a Comparative Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hazem Nour Abdellatif, Assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Hazem nour midline closure
Record Dates: First submitted 2019-10-25; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Midline Incisions; High Risk Patients; Mesh Reinforcement; Incisional Hernia
Keywords: midline reinforcement; incisional hernia; mesh
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Intervention Model Description: two groups one group for onlay mesh position the other for preperitoneal position
Who Masked: Participant
Masking Description: patient don't know the procedure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preperitoneal mesh (Active Comparator): patients underwent preperitoneal mesh mesh placement
  Interventions: Procedure: midline mesh reinforcement
- onlay mesh (Active Comparator): patients underwent preperitoneal mesh mesh placement
  Interventions: Procedure: midline mesh reinforcement

INTERVENTIONS:
Procedure: midline mesh reinforcement — augmentation of midline closure by nonabsorbsble mesh

SUMMARY:
comparison between onlay and preperitoneal augmentation of mid line closure in high risk patients

DETAILED DESCRIPTION:
This study is a randomized comparative clinical trial, carried out in the period from July 2016 to August, 2019, on 47 high-risk patients who are liable to develop incisional hernia, after elective abdominal operations through midline incisions.

High-risk patients means patients who had one or more of the factors that make them more liable to develop incisional hernia, as Obesity, Diabetes mellitus (DM), Steroid therapy, Liver diseases, Renal diseases, Cardiac diseases, Chest diseases , Malignancy, Nutritional deficiency and Old age.

Institutional Review Board, the ethical committee approved the study, determined the number of the study patients, all patients were informed and consented.

Randomization was carried out by assistant nurse using randomization computer program.

The patients were randomly divided into two groups:

* Group I: wound closure is reinforced by onlay polypropylene mesh (24 patients)
* Group II: wound closure is reinforced by preperitoneal polypropylene mesh (23 patients).

In both groups midline laparotomy was closed by non-absorbable continuous suture, 4\1 ratio reinforced with interrupted sutures every 4 bites.

All patients were subjected to: full history taking and clinical examination, radiological and laboratory investigations and endoscopy if needed.

SURGICAL TECHNIQUE In group I patients, after completion of the deemed surgery, the linea alba was closed as mentioned before, then the subcutaneous tissue was dissected of the anterior rectus sheath for 2 cm on both sides, then a polypropylene mesh strip 4 cm width and 4 cm longer than the wound length was applied and centered over the wound, fixed in the onlay position using prolene sutures 2\0. Suction drain is left in position, subcutaneous tissue and skin closed as per usual.

In group II patients, a preperitoneal pocket is created at the time of opening the mid line figure, linea alba is incised separately from peritoneum to facilitate formation of preperitoneal pocket , at time of closure, the mesh was inserted in the preperitoneal space after peritoneal closure with Vicryl 3\0 sutures, the mesh is fixed to the peritoneum by 4 stitches in the 4 quadrants , and to linea alba during midline closure , suction drain was left in the preperitoneal space.

Follow up Patients were followed up in outpatient clinic, (weekly for the first month then monthly for the first six months and lastly every 3 months for one year( in each visit they were carefully examined for any wound occurrences or hernia development, superficial probe ultrasonic examination of abdominal wall was done after 1 week and after 1 month. Demographic data, preoperative, operative and follow up data was collected tabulated and analyzed using SPSS 22 program package.

ELIGIBILITY:
Inclusion Criteria:

* Obesity
* Diabetes mellitus (DM),
* Steroid therapy,
* Liver diseases,
* Renal diseases,
* Cardiac diseases, Chest diseases ,
* Malignancy,
* Nutritional deficiency
* Old age

Exclusion Criteria:

* non risk factor
* previous incisional hernia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
midline incisional hernia , | weekly for one month , then monthly for 6 months then every 3 months later on till one year
  clinical and ultrasound examination of the abdomen for incisional hernia development

SECONDARY OUTCOMES:
post operative complications | (1st month post operative
  hematoma , seroma, wound infection by clinical examination and\or ultrasound

IPD SHARING:
Plan to Share IPD: Undecided